CLINICAL TRIAL: NCT07350642
Title: Efficacy of Platelet Rich Plasma Injection for Vocal Fold Sulcus, Scar and Atrophy
Brief Title: Vocal Fold Injection by Platelet Rich Plasma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Esam Sharkawy, Assistant lecture, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vocal fold injection
Record Dates: First submitted 2025-12-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Vocal Fold Sulcus ,Scar and Atrophy
Keywords: Injection; platelet rich plasma
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with vocal fold scar ,sulcus and atrophy (Other): injection of platelet rich plasma in the vocal fold by special needle
  Interventions: Other: injection of platelet rich plasma; Device: Nasofiberoscopy

INTERVENTIONS:
Other: injection of platelet rich plasma — injection is done percutaneous using a special needle following the guides of surgical anatomy of the neck to reach the area of vocal folds under the effect of local anesthesia and by using nasofiberoscoby
Device: Nasofiberoscopy — It is a type of flexible endoscopies introduced from the patient nose to examine the entire airway reaching the larynx

SUMMARY:
a study to asses safety and efficacy of platelet rich plasma injection in some types of vocal fold problems such as sulcus and atrophy to see the improvement in patient voice and its impact on patient quality of life with a good period of follow up

DETAILED DESCRIPTION:
Vocal fold sulcus, atrophy and scarring are significant causes of dysphonia that present major therapeutic challenges for laryngologists. The etiology of vocal fold scarring is diverse, including phonotrauma, iatrogenic injury from phonomicrosurgery or intubation, malignancy, and radiation therapy. In addition, age-related changes such as the loss of hyaluronic acid, elastic fibers, and bulk causes atrophy can reduce the viable tissue mass.

Vocal fold atrophy leads to reduced pliability and impaired vibratory capacity of the vocal folds. Atrophy is commonly associated with aging (presbyphonia), but it may also result from denervation, disuse, or systemic conditions that affect muscle mass and extracellular matrix composition.

Sulcus vocalis is a structural vocal fold disorder characterized by the presence of a longitudinal furrow along the free edge of the vocal fold. It represents part of the spectrum of SLP disorders, as it involves abnormal thinning, tethering, or loss of the lamina propria, leading to reduced vibratory function. The condition can be congenital, due to defective vocal fold development, or acquired, often associated with chronic inflammation, phonotrauma, or previous vocal fold lesions.

Scarring, atrophy, and sulcus vocalis represent a spectrum of SLP disorders that share pathological features, including inflammatory changes, collagen dysregulation, and depletion of glycosaminoglycans such as hyaluronic acid. Unlike vocal fold paralysis where medialization techniques may restore glottic contact these conditions respond poorly to standard medialization procedures, as glottic gap is not the sole issue. Similarly, exogenous fillers may produce suboptimal vibratory characteristics due to differences in biomechanical properties between artificial materials and native SLP tissue.

These pathological changes primarily affect the superficial lamina propria (SLP) of the vocal folds, an essential layer that provides the viscoelasticity and tensile strength necessary for normal oscillation and sound production.

Disruption of the delicate collagen-elastin-hyaluronic acid balance within the SLP drastically reduces tissue compliance, leading to glottic insufficiency, irregular mucosal wave propagation, and impaired closure. Even minor architectural damage can significantly impact vocal quality, causing dysphonia, vocal fatigue, altered pitch, and decreased quality of life.

Glottic insufficiency due to bowing occurs when the loss of bulk causes the vocal folds to curve inward, leaving a spindle-shaped gap during phonation. This results in increased aperiodicity, as the thin and floppy folds lack sufficient mass and tension for regular vibration. To compensate, patients often engage extrinsic neck muscles to force the folds together, creating hyperfunction that produces a strained, effortful quality and masks the underlying flaccidity.

Current treatment strategies for SLP scarring include voice therapy as a first-line approach, often delivered by specialized speech-language pathologists. In cases with significant glottic insufficiency, surgical augmentation with autologous fat, fascia grafts, or inert injectable materials may be considered; however, these methods carry the risk of further impairing vibratory function. [ Platelet-rich plasma (PRP) has emerged as a promising, minimally invasive alternative. PRP is an autologous concentration of platelets in plasma, enriched with growth factors such as Platelet-erived Growth Factor (PDGF), Vascular Endothelial Growth Factor (VEGF), Transforming Growth Factor-beta (TGF-β), Hepatocyte Growth Facto (HGF), and basic Fibroblast Growth Factor (bFGF), which can stimulate angiogenesis, collagen remodeling, and tissue regeneration.

PRP exerts anti-inflammatory effects by suppressing signaling Nuclear Factor kappa-light-chain-enhancer of activated B cells (NF-κB ) signaling It has been safely applied across multiple fields, including orthopedics, dermatology, plastic surgery, and rheumatology, with low cost and no risk of immune rejection.[6]

ELIGIBILITY:
Inclusion Criteria:

* 1-Age ≥ 10 years 2-Gender: both sexes will be included in the study 3-clinical diagnosis of vocal fold sulcus, scar or atrophy. 4-Diagnosis confirmed by video laryngoscope examination. 5-be able to participate and sign informed consent.

Exclusion Criteria:

1- Laryngeal cancer. 2. Acute laryngeal infection . 3. Systemic diseases that may impair healing, such as:(Uncontrolled diabetes mellitus-Autoimmune disorders affecting the larynx-Coagulopathy or bleeding disorders).

4. Use of systemic corticosteroids or immunosuppressive drugs within the last 4 weeks.

5. Previous laryngeal surgery within the last 6 months 6. Pregnancy or lactation. 7. Known allergy or hypersensitivity to local anesthetics or any component used in PRP preparation.

8. Inability to complete with follow-up visits or voice assessment protocols

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
1-Subjective assessment of the patient using GRBAS scale 2- Subjective assessment of the patien by Arabic version of VHI •3- objective assessment of the patient using video stereoscopic examination and Acoustic analysis • 4-Improvement of patient voice | 4 years
  Arabic version of VHI is a type of questionnaire the smaller score is the better result with a minimum value equal 0 and the maximum one equal 120,viedo stereoscopic examination is done by flexible nasofiberoscopy ,Acoustic analysis is a computerized system to measure different voice parameters ex fundamental frequency ,jitter and shimmer.

CONTACTS AND LOCATIONS:
Overall Officials: Eman sayed hassan sayed eman hassan, professor, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut university, Asyut
  - Faculty of medicine, Asyut

IPD SHARING:
Plan to Share IPD: No